CLINICAL TRIAL: NCT06016296
Title: Effects of Combined Movement and Storytelling Intervention on Fundamental Motor Skills, Language Development and Physical Activity Level in Children Aged 3 to 6 Years: A Randomized Controlled Trial
Brief Title: Combined Movement and Storytelling Intervention on Physical Performance in Children
Acronym: CMSI&Child
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, Academic-Researcher of Department of Physical Activity Sciences, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 105/2021
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Preschool Children
Keywords: Motor Skills; Language Acquisition; Exercise; Preschool; Child
MeSH Terms: conditions — Motor Activity | interventions — Physical Fitness

STUDY DESIGN:
Intervention Model Description: The study includes an experimental design (randomized controlled trial), double-blind, with repeated measures, parallel groups and a quantitative approach.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The assessments will be scheduled two weeks before and after the intervention with a team of evaluators who will not have information about the training groups, nor will the participants know their identities. That is, a double-blind shield
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Upper middle level experimental groups (Experimental): The intervention will be implemented by early childhood educators, who will be previously trained in Combined Movement and Storytelling Intervention (CMSI). Each session will take place in the classroom where the preschoolers usually attend, which will depend on the admission policies of each educational community regarding to level classes (upper middle). The intervention will last 12 weeks (36 sessions), distributed in 3 weekly sessions (Monday, Wednesday and Friday) of 40 minutes per session. The CMSI is based on 2 previous studies, and a book related to CMSI. Twelve unpublished motor stories were elaborated, of which one per week will be executed distributed in 3 sessions per week with the corresponding progressions for each session carried out, placing the children in a sequence of stories that begin with the presentation of a motivating character that will accompany children's in the development of the whole story.
  Interventions: Other: Combined Movement and Storytelling Intervention
- Upper middle level control groups (No Intervention): The upper middle level control groups (n= 2 classes; n= 24 children) will participate in the assessments (initial and final) and will be asked to maintain their regular session of their educational establishments. At the end of the intervention period (according to the results obtained), the control groups children, parents and/or legal guardians, managers and coordinators of each community will be contacted and provided with the material so that they can replicate the experience. In addition, the educators of these establishments (teachers and classroom assistants) will be trained in the CMSI strategy.
- Transition level 1 experimental groups (Experimental): The intervention will be implemented by early childhood educators, who will be previously trained in Combined Movement and Storytelling Intervention (CMSI). Each session will take place in the classroom where the preschoolers usually attend, which will depend on the admission policies of each educational community regarding to level classes (transition level 1). The intervention will last 12 weeks (36 sessions), distributed in 3 weekly sessions (Monday, Wednesday and Friday) of 40 minutes per session. The CMSI is based on 2 previous studies, and a book related to CMSI. Twelve unpublished motor stories were elaborated, of which one per week will be executed distributed in 3 sessions per week with the corresponding progressions for each session carried out, placing the children in a sequence of stories that begin with the presentation of a motivating character that will accompany children's in the development of the whole story.
  Interventions: Other: Combined Movement and Storytelling Intervention
- Transition level 1 control groups (No Intervention): The transition level 1 control groups (n= 2 classes; n= 24 children) will participate in the assessments (initial and final) and will be asked to maintain their regular session of their educational establishments. At the end of the intervention period (according to the results obtained), the control groups children, parents and/or legal guardians, managers and coordinators of each community will be contacted and provided with the material so that they can replicate the experience. In addition, the educators of these establishments (teachers and classroom assistants) will be trained in the CMSI strategy.
- Transition level 2 experimental groups (Experimental): The intervention will be implemented by early childhood educators, who will be previously trained in Combined Movement and Storytelling Intervention (CMSI). Each session will take place in the classroom where the preschoolers usually attend, which will depend on the admission policies of each educational community regarding to level classes (transition level 2). The intervention will last 12 weeks (36 sessions), distributed in 3 weekly sessions (Monday, Wednesday and Friday) of 40 minutes per session. The CMSI is based on 2 previous studies, and a book related to CMSI. Twelve unpublished motor stories were elaborated, of which one per week will be executed distributed in 3 sessions per week with the corresponding progressions for each session carried out, placing the children in a sequence of stories that begin with the presentation of a motivating character that will accompany children's in the development of the whole story.
  Interventions: Other: Combined Movement and Storytelling Intervention
- Transition level 2 control groups (No Intervention): The transition level 2 control groups (n= 2; n= 24 children) will participate in the assessments (initial and final) and will be asked to maintain their regular session of their educational establishments. At the end of the intervention period (according to the results obtained), the control groups children, parents and/or legal guardians, managers and coordinators of each community will be contacted and provided with the material so that they can replicate the experience. In addition, the educators of these establishments (teachers and classroom assistants) will be trained in the CMSI strategy.

INTERVENTIONS:
Other: Combined Movement and Storytelling Intervention — The 40-minute sessions will include three moments: (i) warm-up (5 minutes), which consists of joint mobility exercises and introduction to the motor story of the week; (ii) main part (25 minutes), which incorporates the narration of the motor story by the educator initially, as well as the participation of the children, through their own corporeality with movements based mainly on FMS (locomotion skills and object control) and two way verbal interaction based on questions allusive to the narration delivered by the educator or direct verbal participation cast by each child and; (iii) cool down (10 minutes), where space is provided for the children to gradually return to calm, together with feedback on the contents addressed during the session.
  Other Names: Physical fitness
  Arms: Transition level 1 experimental groups; Transition level 2 experimental groups; Upper middle level experimental groups

SUMMARY:
This study protocol aims to analyze and compare the effects of combined movement and storytelling intervention (CMSI) on fundamental motor skills (locomotor skills and object control), language development (language comprehension, language expression, vocabulary and language description), and physical activity levels (light, moderate to vigorous intensity, and sedentary time) in children aged 3 to 6 years. The sample will consist of 144 children of 12 classes group, randomly assigned to 3 experimental groups (n= 72 children) and 3 control groups (n= 72 children), belonging to 4 classes group of upper middle level classes (2 experimental and 2 control), 4 transition level 1 classes (2 experimental and 2 control) and 4 transition level 2 classes (2 experimental and 2 control). The experimental groups will perform the CMSI for 3 sessions (40-minute per session) per week over 12-weeks (using one motor story per week), while the control groups will not receive any treatment. The main outcome will provide information about fundamental motor skills, language development, and physical activity levels. It is hypothesized that the CMSI has the potential to generate significant increases in selected assessments. If this intervention proves to be beneficial, if could contribute to preschoolers children curricula.

DETAILED DESCRIPTION:
The study includes an experimental design (randomized controlled trial), double-blind, repeated measures and parallel groups (6 interventions and 6 controls) considering previous studies and a quantitative approach. The methodology followed will be the Consolidated Standards of Reporting Trials Statement (CONSORT) methodology.

It is expected to recruit 12 children from each classes group (without distinction of sex). The distribution of the classes groups (12 classes group) will be in 3 experimental groups (6 classes group, n ± 72 children) and 3 control groups (6 classes group, n ± 72 children). The distribution by clusters or strata is justified by the fact that the use of individual randomization would imply a high probability of contaminating the control groups, since it is unfeasible to prohibit children interaction in classrooms or school recreational spaces (i.e., playgrounds, hallways, laboratories), which is where the study intervention will be carried out. The sample size calculation indicates that the ideal number of participants per group is 10. As agreed in a previous study, a mean difference of 3.22 total score of locomotor skills domains was used for this calculation as the minimum difference necessary for substantial clinical relevance, with a standard deviation of 0.70 points, considering an alpha level of 0.05 with a power of 80% and an expected loss of 15%. The GPower program (version 3.1.9.6, Franz Faul, Universiät Kiel, Kiel, Germany) will be used to calculate the statistical power.

The 12 classes group will be selected in 4 upper middle level classes (2 experimental and 2 control; age range between 3 to 4 years), 4 transition level 1 classes (2 experimental and 2 control; age range between 4 to 5 years) and 4 transition level 2 classes (2 experimental and 2 control; age range between 5 to 6 years), which will be randomized by stratified sampling, which consists of segmenting the classes that agreed to participate in the study according to educational levels (strata) and then performing a random sampling on each one of them, using R statistical software, version 4.1.2. This study is considered double-blind because the measurements will be performed by professionals external to the research.

The investigators estimate the participation of 144 children residing in the Maule region, Chile who meet the following inclusion criteria: (i) be enrolled in the educational center (school, college or kindergarten) that commits to participate in the intervention; (ii) age range between 3 to 6 years old; (iii) attend ≥ 85% of the sessions scheduled for the combined movement and storytelling intervention (CMSI). As for the exclusion criteria, will be the following: (i) children with musculoskeletal injuries or medical contraindications (i.e., congenital heart disease, fever, diarrhea or general malaise) that would prevent their normal performance in the assessments and intervention and; (ii) children with permanent educational needs mentioned in Decree Nº83 of the Chilean Ministry of Education, such as, visual, hearing, intellectual or multiple disabilities, dysphasia or autistic disorder.

The current protocol has been reviewed and approved by the Scientific Ethics Committee of the Universidad Católica del Maule, Chile (approval number: N°105/2021, 04 August 2021) and developed following the Declaration of Helsinki for work with human beings.

Before starting the intervention, during the last week of March 2024 (for two weeks), children will be evaluated in the variables considered for the research, later, from the third week of March to the first week of June 2024 (12 weeks) will participate in CMSI. After the intervention (second week of June 2024), for two weeks, the children will undergo the same initial assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in the educational center (school, college or kindergarten) that commits to participate in the intervention.
* Age range between 3 to 6 years old.
* Attend ≥ 85% of the sessions scheduled for the CMSI.

Exclusion Criteria:

* Children with musculoskeletal injuries or medical contraindications (i.e., congenital heart disease, fever, diarrhea or general malaise) that would prevent their normal performance in the assessments and intervention.
* Children with permanent educational needs mentioned in Decree Nº83 of the Chilean Ministry of Education, such as, visual, hearing, intellectual or multiple disabilities, dysphasia or autistic disorder.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from fundamental Motor Skills | 2 weeks
  It will be assessed by means of the test of gross motor development-second edition (TGMD-2). This battery measures 12 fundamental motor skilss in two different domains (locomotor skills and object control), the locomotor skills domain contains 6 assessments: (i) running, (ii) galloping, (iii) hopping on one foot, (iv) long jumping, (v) horizontal jumping and, (vi) lateral sliding. The object control domain also includes 6 assessments: (i) batting a stationary ball, (ii) stationary dribbling, (iii) catching a ball, (iv) kicking a ball, (v) throwing a ball and, (vi) rolling a ball. Estimated administration time is ≤ 10 minutes per children. The 6 locomotion skills and 6 object control include 24 criteria, allowing a total score from 0 to 48 points. The higher score, better FMS.
Change from language development | 2 weeks
  The language test for preschoolers (TELEPRE), will be used. The purpose of this assessment is to measure the language of children in initial educational levels (3 to 6 years old) by means of 4 domains: (i) language comprehension, (ii) language expression, (iii) vocabulary and, (iv) language description. The administration of the instrument requires a booklet of questions, some objects (bottle, toy car, pencil, plate, needle, cup, paintbrush, screw, sponge, small ball, button, small book, spoon, scissors, matchbox; plus, three objects that serve as distractors) and 3 representative pictures of situations (i.e., serving milk to a cat, setting the table and being in a toy store) to be described by the child. To administer the instrument, a room free of disturbing noises is required, in which the evaluator, the child and a classroom assistant will be present. The estimated application time is ≤ 25 minutes. The higher score, better language development.
Change from physical activity level | 2 weeks
  It will be objectively monitored by accelerometers (ActiGraph GT9X, Pensacola, FL, USA). The device will be worn at the waist on an elastic belt, at the mid-axillary line on the right side. Children will be instructed to wear the accelerometer 24 hours a day, for at least 7 days, including 2 weekend days, and only removed the device when bathing or engaged in water activities. The minimum amount of data considered acceptable for analysis purposes will be 5 days (including one weekend day), with at least 10 hours/day of wear time. Light, moderate to vigorous intensity, and sedentary time will be considered to analysis, while sleep time will be not taken into account. Data will be verified using Actilife software version 5.6 (ActiGraph, Pensacola, FL, USA). Consecutive 20-min blocks of 0 count will considered as non-use of the device and discarded from the analyses.

SECONDARY OUTCOMES:
Bipedal height | 2 weeks
  Will be measured by placing a tape measure (Bodymeter 206, SECA, Germany; accuracy of 0.1 cm) on the wall and utilizing the Frankfort plane in a horizontal position (assessment in cm).
Circumferences and skinfolds | 2 weeks
  Will be measured with an inextensible tape measure (Seca-201, Germany) with an accuracy of 0.1 cm. Similarly, skinfolds (mm) measured in the bicipital, tricipital, subscapular and suprailiac regions will be measured using a plicometer (Harpenden-FG1056, England; accuracy of 0.2 mm) that exerts a constant pressure of 10 g/mm2.
Sociodemographic Variables | 2 weeks
  Legal guardians will be asked to respond to the following: (i) child's name; (ii) child's date of birth; (iii) in which country the child was born; (iv) in which country was I born; (v) what is my family relationship to the child; (vi) marital status of the parents or guardians; (vii) in what area does the child reside; (viii) the place where the child lives has a yard; (ix) how many people live with the child; (x) how many persons work in participants household; (xi) what is the total family income of the people living with the child (approximately); (xii) what is the highest level of schooling participant have.
Body weight | 2 weeks
  Will be determined using an electronic scale (Tanita BC-730 Tokyo, Japan; accuracy of 0.1 kg) in kg.
Body mass index | 2 weeks
  Will be computed by dividing the body weight by the square of the bipedal height (kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Valdés-Badilla, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Poliderportivo San Clemente, San Clemente, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared. The investigators will only disseminate the results of the study through scientific papers and presentations at scientific congresses.

REFERENCES:
- [Result] Willumsen J, Bull F. Development of WHO Guidelines on Physical Activity, Sedentary Behavior, and Sleep for Children Less Than 5 Years of Age. J Phys Act Health. 2020 Jan 1;17(1):96-100. doi: 10.1123/jpah.2019-0457. PMID 31877559
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] den Uil AR, Janssen M, Busch V, Kat IT, Scholte RHJ. The relationships between children's motor competence, physical activity, perceived motor competence, physical fitness and weight status in relation to age. PLoS One. 2023 Apr 14;18(4):e0278438. doi: 10.1371/journal.pone.0278438. eCollection 2023. PMID 37058506
- [Result] Ma FF, Luo DM. Relationships between physical activity, fundamental motor skills, and body mass index in preschool children. Front Public Health. 2023 Apr 12;11:1094168. doi: 10.3389/fpubh.2023.1094168. eCollection 2023. PMID 37124831
- [Result] Duncan MJ, Hall C, Eyre E, Barnett LM, James RS. Pre-schoolers fundamental movement skills predict BMI, physical activity, and sedentary behavior: A longitudinal study. Scand J Med Sci Sports. 2021 Apr;31 Suppl 1:8-14. doi: 10.1111/sms.13746. PMID 33871088
- [Result] Webster EK, Sur I, Stevens A, Robinson LE. Associations between body composition and fundamental motor skill competency in children. BMC Pediatr. 2021 Oct 11;21(1):444. doi: 10.1186/s12887-021-02912-9. PMID 34629074
- [Result] Bolger LE, Bolger LA, O'Neill C, Coughlan E, O'Brien W, Lacey S, Burns C, Bardid F. Global levels of fundamental motor skills in children: A systematic review. J Sports Sci. 2021 Apr;39(7):717-753. doi: 10.1080/02640414.2020.1841405. Epub 2020 Dec 30. PMID 33377417
- [Result] Mule D, Jeger I, Dotsch J, Breido F, Ferrari N, Joisten C. Correlation between Language Development and Motor Skills, Physical Activity, and Leisure Time Behaviour in Preschool-Aged Children. Children (Basel). 2022 Mar 18;9(3):431. doi: 10.3390/children9030431. PMID 35327803
- [Result] Lin J, Zhang R, Shen J, Zhou A. Effects of school-based neuromuscular training on fundamental movement skills and physical fitness in children: a systematic review. PeerJ. 2022 Jul 8;10:e13726. doi: 10.7717/peerj.13726. eCollection 2022. PMID 35833011
- [Result] Van Capelle A, Broderick CR, van Doorn N, E Ward R, Parmenter BJ. Interventions to improve fundamental motor skills in pre-school aged children: A systematic review and meta-analysis. J Sci Med Sport. 2017 Jul;20(7):658-666. doi: 10.1016/j.jsams.2016.11.008. Epub 2017 Jan 23. PMID 28169146
- [Result] Han X, Zhao M, Kong Z, Xie J. Association between fundamental motor skills and executive function in preschool children: A cross-sectional study. Front Psychol. 2022 Aug 25;13:978994. doi: 10.3389/fpsyg.2022.978994. eCollection 2022. PMID 36092056
- [Result] Jylanki P, Mbay T, Hakkarainen A, Saakslahti A, Aunio P. The effects of motor skill and physical activity interventions on preschoolers' cognitive and academic skills: A systematic review. Prev Med. 2022 Feb;155:106948. doi: 10.1016/j.ypmed.2021.106948. Epub 2021 Dec 30. PMID 34974071
- [Result] Eyre ELJ, Clark CCT, Tallis J, Hodson D, Lowton-Smith S, Nelson C, Noon M, Duncan MJ. The Effects of Combined Movement and Storytelling Intervention on Motor Skills in South Asian and White Children Aged 5-6 Years Living in the United Kingdom. Int J Environ Res Public Health. 2020 May 13;17(10):3391. doi: 10.3390/ijerph17103391. PMID 32414027
- [Result] Turner L, Shamseer L, Altman DG, Weeks L, Peters J, Kober T, Dias S, Schulz KF, Plint AC, Moher D. Consolidated standards of reporting trials (CONSORT) and the completeness of reporting of randomised controlled trials (RCTs) published in medical journals. Cochrane Database Syst Rev. 2012 Nov 14;11(11):MR000030. doi: 10.1002/14651858.MR000030.pub2. PMID 23152285
- [Result] Parker K, Nunns MP, Xiao Z, Ford T, Ukoumunne OC. Characteristics and practices of school-based cluster randomised controlled trials for improving health outcomes in pupils in the UK: a systematic review protocol. BMJ Open. 2021 Feb 15;11(2):e044143. doi: 10.1136/bmjopen-2020-044143. PMID 33589463
- [Result] Manacero S, Nunes ML. Longitudinal study of sleep behavior and motor development in low-birth-weight preterm children from infancy to preschool years. J Pediatr (Rio J). 2021 Jan-Feb;97(1):44-51. doi: 10.1016/j.jped.2019.10.010. Epub 2020 Feb 20. PMID 32088142
- [Result] Cano-Cappellacci M, Leyton FA, Carreno JD. Content validity and reliability of test of gross motor development in Chilean children. Rev Saude Publica. 2015;49:97. doi: 10.1590/S0034-8910.2015049005724. Epub 2015 Dec 31. PMID 26815160
- [Result] Valentini NC. Validity and reliability of the TGMD-2 for Brazilian children. J Mot Behav. 2012;44(4):275-80. doi: 10.1080/00222895.2012.700967. Epub 2012 Aug 2. PMID 22857518
- [Result] Kim S, Kim MJ, Valentini NC, Clark JE. Validity and reliability of the TGMD-2 for South Korean children. J Mot Behav. 2014;46(5):351-6. doi: 10.1080/00222895.2014.914886. Epub 2014 Jun 10. PMID 24915525
- [Result] Estivaleti JMO, Bergamo RR, Oliveira LC, Beltran DCG, Silva Junior JPD, Santos MD, Matsudo VKR. Physical activity level measured by accelerometry and physical fitness of schoolchildren. Rev Paul Pediatr. 2022 Sep 9;41:e2021230. doi: 10.1590/1984-0462/2023/41/2021230. eCollection 2022. PMID 36102399
- [Result] Migueles JH, Cadenas-Sanchez C, Ekelund U, Delisle Nystrom C, Mora-Gonzalez J, Lof M, Labayen I, Ruiz JR, Ortega FB. Accelerometer Data Collection and Processing Criteria to Assess Physical Activity and Other Outcomes: A Systematic Review and Practical Considerations. Sports Med. 2017 Sep;47(9):1821-1845. doi: 10.1007/s40279-017-0716-0. PMID 28303543
- [Result] Kuzik N, Naylor PJ, Spence JC, Carson V. Movement behaviours and physical, cognitive, and social-emotional development in preschool-aged children: Cross-sectional associations using compositional analyses. PLoS One. 2020 Aug 18;15(8):e0237945. doi: 10.1371/journal.pone.0237945. eCollection 2020. PMID 32810172
- [Result] Robinson LE, Stodden DF, Barnett LM, Lopes VP, Logan SW, Rodrigues LP, D'Hondt E. Motor Competence and its Effect on Positive Developmental Trajectories of Health. Sports Med. 2015 Sep;45(9):1273-1284. doi: 10.1007/s40279-015-0351-6. PMID 26201678
- [Result] Logan SW, Ross SM, Chee K, Stodden DF, Robinson LE. Fundamental motor skills: A systematic review of terminology. J Sports Sci. 2018 Apr;36(7):781-796. doi: 10.1080/02640414.2017.1340660. Epub 2017 Jun 21. PMID 28636423
- [Result] Lyster SH, Lervag AO, Hulme C. Preschool morphological training produces long-term improvements in reading comprehension. Read Writ. 2016;29:1269-1288. doi: 10.1007/s11145-016-9636-x. Epub 2016 Mar 17. PMID 27340335
- See also: Chilean Ministry of Education. Diversificacion de la enseñanza — https://especial.mineduc.cl/wp-content/uploads/sites/31/2016/08/Decreto-83-2015.pdf
- See also: Test of gross motor development-2 — https://33202576.weebly.com/uploads/1/4/6/8/14680198/tgmd-2-2.pdf
- See also: Prueba de Desarrollo del Lenguaje para Pre-Escolares TELEPRE 1 — https://es.scribd.com/document/76165919/Prueba-TELEPRE